CLINICAL TRIAL: NCT07190976
Title: The Value of EEG in Stroke Units
Status: Recruiting | Type: Observational
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, Panagiota Eleni Tsalouchidou, Dr. med. Panagiota Eleni Tsalouchidou, Attikon Hospital
Other Study IDs: 48827/27.05.2024
Record Dates: First submitted 2025-09-17; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients with acute ischemic or hemorrhagic stroke
  Interventions: Other: Routine EEG

INTERVENTIONS:
Other: Routine EEG — The study is observational. No intervention is anticipated. Patients will be submitted to EEG recording within the first seven days of stroke
Other: Routine EEG — The study is observational

SUMMARY:
Τhe aim of the study is to investigate the role of EEG both in predicting epileptogenesis in patients with acute stroke and in detecting and clarifying the clinical significance of subclinical epileptic seizures in a stroke unit. More specifically, the performance of routine EEG in patients with ischemic or hemorrhagic stroke who are hospitalized in the Stroke Unit within the first days after the event, regardless of the presence of clinical indications, and the identification of risk factors for the early development of epilepsy in the course of these patients' disease constitute the central research question. The identification of patients with subclinical electroencephalographic seizures and the impact of such events on functional outcome, as well as their association with the development of epilepsy, are set as secondary research objectives.

ELIGIBILITY:
Inclusion Criteria: Patients over 18 years of age with confirmed acute ischemic or hemorrhagic stroke are eligible for inclusion in the study. Patients whose clinical presentation mimics that of a stroke will be included until the diagnosis of stroke is ruled out, at which point they will be excluded from the study.

-

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with acute ischemic or hemorrhagic stroke in whom it is not possible to perform an electroencephalogram within the first 7 days after the event, as well as patients who themselves or their legal representatives do not consent to participation, will be excluded from the study.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of post-stroke epilepsy | 4 years

CONTACTS AND LOCATIONS:
Locations (1):
- University General Hospital "ATTIKON"- General Hospital of West Attica "H AGIA VARVARA" 2nd Neurology Clinic, NKUA, Chaïdári, Athens, Greece